CLINICAL TRIAL: NCT05628298
Title: Pulsed Heat as a Drug-free Treatment for Pregnancy Related Pain
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Soovu Labs Inc. (Industry)
Collaborators: Virginia Mason Hospital/Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: R23-22
Record Dates: First submitted 2022-11-16; First posted 2022-11-28 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Pain; Pain, Labor
Keywords: pain; pregnancy; Female
MeSH Terms: conditions — Pain; Labor Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Experimental group: Women in their 2nd and 3rd trimester of pregnancy who have significant pregnancy related pain (>5/10). Subjects will be allowed to use the device during labor and one month postpartum.
  Interventions: Device: Soovu Pain Relief System

INTERVENTIONS:
Device: Soovu Pain Relief System — The Soovu Pain Relief system uses pulses of heat to block the TRPV-1 calcium channel on peripheral pain nerves. The study will determine if the FDA cleared device significantly reduces the subject's pregnancy related pain.

SUMMARY:
Studies indicate that up to 75% of women will experience pain sometime during their pregnancy. Recent recommendations by the FDA recommended that non-steroidal anti-inflammatory (NSAIDS) medications be avoided during pregnancy. This recommendation limits the pain medications available for use during pregnancy.

Antidotal evidence suggests that the FDA cleared Soovu pulsed heat device may produce pain relief during pregnancy. This study tests the Soovu device's ability to provide pain relief during pregnancy and up to one month post-partum and may eventually offer a safe nondrug option to treat pregnancy related pain.

This is an observational pilot study

The primary objective and hypothesis of this study is that the use of the Soovu pain management device will produce a significant reduction of pain when comparing pre versus post treatment pain.

DETAILED DESCRIPTION:
Pain associated with pregnancy occurs in approximately 60 to 70% of women. The mechanism of action of pulsed heat and TRPV-1 blockade is expected to be relevant in this population based on the etiology of their pain, and should help reduce their pain. In addition, there have been several pregnant women who have used the device to treat their pain associated with pregnancy. Their use was driven partly based on the FDA's recommendation to avoid non-steroidal anti-inflammatory medications limiting medication options. Based on these antidotal experiences and feedback, as well as the device's mechanism of action, this study is proposed.

The study is a pilot observational study that will provide results to support a larger more rigorous and involved clinical trial.

1. The primary objective of this study is to determine whether the Soovu Pain Relief device is effective in reducing pain associated with pregnancy in the 2nd and 3rd trimester and in the first month postpartum.
2. The secondary objectives include testing whether the study device reduces the effects of pain on physical function and the satisfaction and opinions of both subjects and providers on the effectiveness and usability of the study device. Subjects will also be asked about and needed pain medication use and their experience with the device if they used it during delivery.

Study design This is a single center nonrandomized non blinded pilot study on the effects of the Soovu Pain Relief device in pregnancy associated pain. 25-35 subjects are planned in the study which covers the 2nd and 3rd trimester and one month post-partum. Subjects will be referred to the study by their care providers or via posters in the clinic. Each subject who enters the study will receive a Soovu Pain Relief device with instructions on its use. All subjects will continue to receive their usual care. There are no visits associated with involvement in the study. Subjects can elect to use the device to treat their pain during the study and will record their pain level pre and post use. The data is collected via the phone app that controls the device. Screening data will be reviewed to determine subject eligibility. Subjects who meet all inclusion criteria and none of the exclusion criteria will be entered into the study.

The total duration of the study is expected to be 14 months. 6-7 months for subject recruitment and 7 months for final subject follow-up.

The primary efficacy endpoint is the difference between the numerical pain score (0-10) pretreatment versus post treatment. Pain relief is the primary outcome measure as related to the study pain management device.

Secondary Efficacy Endpoints The secondary efficacy endpoints include whether the study device reduces the effects of pain on physical function and the satisfaction and opinions of both subjects and providers on the effectiveness and usability of the study device. The physical function questionnaire is a well validated instrument form the PROMIS outcome library and is a measure of function not necessarily pain. The usability and satisfaction evaluations help determine subject and provider acceptance of the device and can lead to product improvements.

The primary outcomes measure is pain level pre versus post treatment with the Soovu Device on a 0-10 point numeric scale. The data will be modeled as a repeated measures ordinal regression (primary choice), or a repeated measures model on a continuous response.

Analysis of Secondary Endpoints Changes on the PROMIS pain interference short form measure given on a monthly basis during the study will be analyzed using a Anova repeated measures technique.

Subject satisfaction with the experimental Soovu device at monthly intervals and one month post-partum if indicated (Likert scale) will be tabulated and represented as a mean value with standard deviations. Subjects will also be asked whether they needed any supplemental pain medications and the name or type of medications.

Provider assessment and opinions of device (Likert scale) at study conclusion and one month post-partum. The results will be tabulated and represented as a mean value with standard deviations.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant subjects in the second and third trimester of pregnancy with pain related to their pregnancy.
2. Subjects must have a pain level greater then 4 on a 0-10 point numeric pain scale.
3. Subjects between the ages of 18 and 60 years old.
4. Written informed consent obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

1. Subjects felt to have any condition or complication related to their pregnancy that their provider recommends that the subject abstains from the use of the Soovu device.
2. Subjects with a BMI > 0.45
3. Subjects who have a significant ongoing pain problem unrelated to their pregnancy that would make interpretation of their study data uncertain.
4. Presence of a condition or abnormality that in the opinion of the investigator or provider would compromise the safety of the patient or the quality of the data.

Ages: 18 Years to 60 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Pregnant females
Study Population: Pregnant females in their 2nd and third trimester with pregnancy related pain
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2023-01-15 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Changes in pain level | After each treatment over a six month period
  Changes in pain level before and after treatment as measured by PROMIS NPR

SECONDARY OUTCOMES:
Changes in pain interference scale | Monthly over six months
  • Changes on the PROMIS pain interference short form measure given on a monthly basis during the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Virginia Mason Medical center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No